CLINICAL TRIAL: NCT03893656
Title: Retroperitoneoscopic Donor Nephrectomy: a Retrospective Single-center Study
Brief Title: Retroperitoneoscopic Donor Nephrectomy
Acronym: RDN
Status: Completed | Type: Observational
Sponsor: Samsun Liv Hospital (Other)
Collaborators: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Mehmet Necmettin Mercimek, Principal investigator, MD, Samsun Liv Hospital
Other Study IDs: OMU KAEK (2019/79)
Record Dates: First submitted 2019-03-24; First posted 2019-03-28 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Transplant; Complication, Failure
Keywords: Living donor nephrectomy; Kindey transplantation; Retroperitoneoscopic donor nephrectomy; Hernia
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
to compare the results of right and left-sided retroperitoneoscopic donor nephrectomy (RDN).

DETAILED DESCRIPTION:
This was a retrospective study evaluating demographics, intraoperative and postoperative data of 158 kidney donors who underwent RDN from January 2010 to August 2018. Two groups were created according to the side of the surgery including Right RDN (group 1) and left RDN (group 2). The results of the recipients' were also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Adult donors
* Kidney donors undergoing retroperitoneoscopic donor nephrectomy
* Recipients of the kidneys
* Donors with the consent form
* Recipients with consent form

Exclusion Criteria:

* open donor nephrectomies
* donors without the consent form
* Recipients without the consent form

Ages: 18 Years to 57 Years | Sex: All
Age Groups: Adult
Study Population: 158 consecutive kidney donors undergoing pure RDN for allotransplantation at Ondokuz Mayıs University from January 2010 to August 2018. All operations were performed by a single surgeon (E. O.).
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2019-05-08 (Actual); Study Completion 2019-07-22 (Actual)

PRIMARY OUTCOMES:
Operation time | at the end of the surgery
  time from onset to complete of surgery
Blood loss | at the end of the surgery
  amount of bleeding during surgery (mililiter)
warm ishemia time | at the end of the surgery
  time from renal artery and vein dissection of the kidney to the initiation of perfusion on the bench table.
İntraoperative complications | at the end of the surgery
  abnormal problems that may be seen during surgery and require additional intervention.
incisional hernia | up to 2 years
  abdominal incision or trocar site defects of donors
postoperative complication | up to 1 month
  abnormal problems that may be seen after surgery and require additional intervention or follow-up (grade I-V)

CONTACTS AND LOCATIONS:
Overall Officials: Saban Sarıkaya, Professor, Study Chair — Ondokuz Mayıs University
Locations (2):
- Turkey (Türkiye) (2):
  - Samsun Liv Hospital, Samsun
  - Ondokuz Mayıs University, Samsun

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Result] Ratner LE, Ciseck LJ, Moore RG, Cigarroa FG, Kaufman HS, Kavoussi LR. Laparoscopic live donor nephrectomy. Transplantation. 1995 Nov 15;60(9):1047-9. PMID 7491680
- [Result] Hsu JW, Reese PP, Naji A, Levine MH, Abt PL. Increased early graft failure in right-sided living donor nephrectomy. Transplantation. 2011 Jan 15;91(1):108-14. doi: 10.1097/TP.0b013e3181fd0179. PMID 21441855
- [Result] Kumar A, Chaturvedi S, Gulia A, Maheshwari R, Dassi V, Desai P. Laparoscopic Live Donor Nephrectomy: Comparison of Outcomes Right Versus Left. Transplant Proc. 2018 Oct;50(8):2327-2332. doi: 10.1016/j.transproceed.2018.03.034. Epub 2018 Mar 16. PMID 30316352